CLINICAL TRIAL: NCT00536614
Title: A Randomized Phase II Study of Gemcitabine/Cisplatin With or Without Cetuximab to Evaluate the Efficacy in Patients With Locally Advanced or Metastatic EGFR-EGFR-Positive Pancreatic Cancer. SpaCe Trial
Brief Title: Gemcitabine/Cisplatin +/-Cetuximab in Patients With Locally Advanced or Metastatic EGFR-Positive Pancreatic Cancer
Acronym: SPaCe-01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano per lo studio dei Carcinomi dell'Apparato Digerente (Other)
Collaborators: Mario Negri Institute for Pharmacological Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-004309-69
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Last update posted 2007-09-28 (Estimated); Status verified 2007-09

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; metastatic; EGFR; locally advanced pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (No Intervention): arm A) gemcitabine/cisplatin in combination with Cetuximab arm B) gemcitabine/cisplatin alone
  Interventions: Genetic: cetuximab

INTERVENTIONS:
Genetic: cetuximab — Cetuximab is an EGFR antibody inhibitor; it has been shown to increase the activity of gemcitabine (GEM) in advanced pancreatic cancer.

SUMMARY:
This is multicenter, open-label, randomized, phase II trial in patients with locally advanced or metastatic pancreatic cancer. Primary objective: objective response rate. Secondary objectives: safety, time to disease progression, median duration of response, time to treatment failure, overall survival time, correlation between bio-pathological characterization (EGFR, akt, MAPks) objective response and survival

DETAILED DESCRIPTION:
During the last years, the esocrine pancreatic carcinoma presented a slow but constant increase of incidence. Chemotherapy determined disappointing results. Gemcitabine determined a slight advantage in survival and clinical benefit in comparison with gemcitabine with cisplatin or oxaliplatin Elevated expression of EGFR or its ligand correlates with worse prognosis in a variety of human cancers including pancreatic cancer. Therefore, blockade of EGFR activity would provide a novel strategy for the treatment of cancer. Cetuximab (C225) is a human/murine chimeric monoclonal antibody directed to the EGFR binding site. In a preclinical setting, Cetuximab has demonstrated anticancer activity both in cell culture experiments and in "in vivo" tumor xenograft animal model Since the combination of gemcitabine and cisplatin seems to be the more effective treatment for advanced pancreatic cancer and Cetuximab may improve activity of this combination we designed this phase II randomised trial to assess the role of Cetuximab in combination with gemcitabine and cisplatin in pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically confirmed diagnosis of adenocarcinoma of the pancreas
* Locally advanced (non-resectable) or metastatic pancreatic cancer
* Presence of at least one uni-dimensional indicator lesion measurable by CT scan or MRI in not an irradiated area (RECIST criteria)
* Immunohistochemical evidence or positive EGFR expression prior to study entry in primary tumor and/or at least one metastasis
* Life expectancy of ≥ 3 months
* Karnofsky performance status of ≥70 at study entry
* Neutrophils ≥ 1.5 x 109/L, platelets ≥100 x 109/L, and hemoglobin ≥ 9 g/dL
* Bilirubin level either normal or < 1.5 x ULN
* ASAT and ALAT ≤ 2.5 X ULN (≤ 5 x ULN if liver metastasis are present)
* Serum creatinine < 1.5 x ULN
* Effective contraception for both, male and female patients if the risk of conception exists
* Signed written informed consents prior to beginning protocol specific procedures

Exclusion Criteria:

* Brain metastasis
* Previous chemotherapy for locally advanced or metastatic pancreatic cancer
* Adjuvant therapy is allowed if recurrence is documented > 6 months after the end of adjuvant treatment
* Radiotherapy within 4 weeks prior to study entry
* Concurrent chronic systemic immune therapy
* Any investigational agent(s) 4 weeks prior to entry
* Previous exposure to EGF, monoclonal antibodies, signal transduction inhibitors or EGFR targeting therapy
* Clinically relevant coronary artery disease or a history of a myocardial infarction within the last 12 months
* Known grade 3 or 4 allergic reaction to any of the components of the treatment
* Known drug abuse/ alcohol abuse
* Legal incapacity or limited legal capacity
* Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent
* Women who are pregnant or breastfeeding
* Any concurrent malignancy other than non-melanoma skin cancer, or carcinoma in situ of the cervix. (Patients with a previous malignancy but without evidence of disease for ≥ 5 years will be allowed to enter the trial).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2005-05; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Overall survival | A subject's survival time will be defined as the time from randomization to the date of his or her death. If the subject has not died, survival will be censored on last date the subject was known to be alive.

SECONDARY OUTCOMES:
response to treatment, and toxicity | the time from randomization until the date of discontinuation of treatment or progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Cascinu, MD, Study Chair — Gruppo Italiano per lo studio dei Carcinomi dell'Apparato Digerente
Locations (10):
- Italy (10):
  - A.O. Ospedale Umberto I - Università - Località Torretta, Ancona, Ancona
  - Ospedali Riuniti, Largo Barozzi, 1, Bergamo, Bergamo
  - A.O. Treviglio-Caravaggio, P.le Ospedale n1, Treviglio, Bergamo
  - Casa di Cura di Poliambulanza, Via Bissolati 57, Brescia, Brescia
  - A.O. Careggi-Università, Viale Pieraccini, 17, Florence, Firenze
  - Azienda USL 6 - Viale Alfieri, 36, Livorno, Livorno
  - A.O. Carlo Poma - Via Albertoni, 1, Mantova, Mantova
  - A.O. Cà Granda, Piazza Ospedale Maggiore, 3, Milan, Milano
  - Ospedale S.Gerardo, Via Donizetti, 106, Monza, Milano
  - Università Campus Biomedico, Via Emilio Longoni, 83, Roma, Roma

REFERENCES:
- [Derived] Cascinu S, Berardi R, Labianca R, Siena S, Falcone A, Aitini E, Barni S, Di Costanzo F, Dapretto E, Tonini G, Pierantoni C, Artale S, Rota S, Floriani I, Scartozzi M, Zaniboni A; Italian Group for the Study of Digestive Tract Cancer (GISCAD). Cetuximab plus gemcitabine and cisplatin compared with gemcitabine and cisplatin alone in patients with advanced pancreatic cancer: a randomised, multicentre, phase II trial. Lancet Oncol. 2008 Jan;9(1):39-44. doi: 10.1016/S1470-2045(07)70383-2. PMID 18077217